CLINICAL TRIAL: NCT00983541
Title: Definitive Chemoradiation With Gemcitabine and Continuous 5- FU (Fluorouracil)Followed by High Dose Rate Brachytherapy or Stereotactic Body Radiation Therapy Boost in Locally Advanced Intra or Extrahepatic Cholangiocarcinoma
Brief Title: Chemoradiation +Gemcitabine +Continuous 5-FU (Fluorouracil) Followed by High Dose Brachytherapy/Stereotactic Radiation Boost in Locally Advanced Intra/Extrahepatic Cholangiocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI35306
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-07

CONDITIONS: Cancer
Keywords: intra or extrahepatic cholangiocarcinoma; liver cancer; liver; HCC; EHCC
MeSH Terms: conditions — Neoplasms; Cholangiocarcinoma; Liver Neoplasms | interventions — Fluorouracil; Brachytherapy; Radiosurgery; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Fluorouracil (5-FU); Radiation: Brachytherapy or SBRT (Stereotactic body radiation therapy); Drug: Gemcitabine

INTERVENTIONS:
Drug: Fluorouracil (5-FU) — 5-FU Injection,USP (GeneraMedix Inc.) is effective in palliative management of carcinoma (colon, rectum, breast, stomach, pancreas) FDA approved in 1962-NDA (New Drug Application)012209. This study uses 350 mg/m2/day days 1-5 each week of radiation therapy
  Other Names: (5-FU)
Radiation: Brachytherapy or SBRT (Stereotactic body radiation therapy) — Patients receive 45 Gy (gray) external beam radiation therapy including the primary tumor and regular lymph nodes (25 fractions over 5 weeks). Within 1 month of external beam radiation therapy, patients will have boost treatment of 20 Gy in 4 fractions, via Ir-192 brachytherapy or SBRT (Stereotactic Body Radiation Therapy).
  Other Names: brachytherapy or stereotactic body radiation therapy boost
Drug: Gemcitabine — Pancreatic:Indicated as first line treatment for patients with locally advanced (nonresectable Stage II or III) or metastatic(Stage IV) pancreatic adenocarcinoma.
  Ovarian:Gemzar with carboplatin is indicated for treatment of patients with advanced ovarian cancer relapsed 6 months after plat-based therapy.
  Breast:Gemzar with paclitaxel is indicated for first line treatment of patients with metastatic breast cancer after failed anthracycline-containing adjuvant chemotherapy, unless anthracyclines.
  Non-small cell lung cancer(NSCLC):Gemzar is indicated with cisplatin for first line treatment of patients with inoperable, local advanced (Stage IIIA/IIIB), metastatic (Stage IV) NSCLC.
  Other Names: Gemzar

SUMMARY:
OBJECTIVES: This study proposes to evaluate the feasibility of delivery of this treatment in terms of toxicity. If toxicity is not acceptable, the treatment is not feasible.

Primary Objectives

* To establish a preliminary assessment whether toxicity rates are acceptable in patients with locally advanced intra or extrahepatic cholangiocarcinoma when treated with a regimen of gemcitabine every two weeks and continuous fluorouracil (5-FU) given concurrently with external beam radiation therapy to a total dose of 45 gray(Gy), followed by a brachytherapy or Stereotactic Body Radiation Therapy(SBRT) boost.

Secondary Objectives

* To evaluate the overall survival rate, progression free survival rate, tumor response rate, local control rate and the rate of distant metastases following gemcitabine and continuous 5-FU concurrent with radiation therapy in patients with locally advanced intra or extrahepatic cholangiocarcinoma.
* To evaluate the rate at which patients with unresectable extrahepatic cholangiocarcinoma become resectable following gemcitabine and radiation therapy.

DETAILED DESCRIPTION:
Cholangiocarcinoma is an uncommon tumor arising from the biliary tract. It can be stratified into two categories based on location, intrahepatic and extrahepatic. In the United States, approximately 4,000-5,000 cases of cholangiocarcinoma are diagnosed each year. The most common location is at the bifurcation of the common hepatic duct and is classified as extrahepatic, also known as a Klatskin tumor. Approximately 60-80% of tumors are found in this perihilar location. A history of primary sclerosing cholangitis confers 10% lifetime risk of developing cholangiocarcinoma. Other known risk factors include ulcerative colitis, liver fluke infestations, hepatolithiasis, thorotrast exposure and choledochal cysts. Cholecystectomy decreases the risk. Most patients are lymph node positive at diagnosis, approaching 55-60%, and less than half are resectable at diagnosis.

Because of the rare nature of the tumor, there are limited prospective trials addressing the roles for surgery, chemotherapy (CT) and radiation therapy (RT) in the treatment of cholangiocarcinoma. Despite advances in surgical and radiotherapy techniques, the prognosis for cholangiocarcinoma remains dismal. Historically, survival is poor with a 0-10% 5-year survival. In more recent years, a median survival of 2-15 months is expected. Patients who are able to undergo surgical resection at diagnosis have longer survival of approximately 20-24 months. Recent investigations in the area of neoadjuvant chemoradiation followed by orthotopic liver transplant in a select group of patients report promising results, with 1-, 3- and 5-year overall survival of 92%, 82% and 82%, respectively. Although this approach may be appropriate for select patients, namely younger patients with small tumors, no or limited nodal involvement, and no encasement of the major vasculature, the majority of patients presenting with cholangiocarcinoma will present with unresectable disease at initial diagnosis, often due to nodal involvement.

Chemotherapy The role of chemotherapy (CT) in cholangiocarcinoma has not been established. Most chemotherapy trials have been small single institution phase II trials, and there have been no large prospective randomized trials. Additionally, most chemotherapy trials include patients with intrahepatic, extrahepatic and gallbladder carcinomas, as well as patients with locally advanced and metastatic disease. Response rates have ranged from 0-40% with no complete remissions. The most extensively investigated CT agent has been 5-fluorouracil (5-FU), which has disappointing response rates of 9% as a single agent. Response rates were not improved by the addition of streptozotocin or methyl-CCNU (Semustine) to 5-FU in a randomized trial performed by Eastern Cooperative Oncology Group (ECOG).6 Multiple combination CT regimens have been investigated in small clinical trials, and none have shown a survival benefit.

Gemcitabine has shown some promise as a potential chemotherapeutic agent in the treatment of cholangiocarcinoma. A multicenter retrospective analysis out of Japan examining a multitude of different CT regimens in patients with intrahepatic, extrahepatic or gallbladder carcinomas reported gemcitabine was the most effective treatment, with a reduction in mortality by about 50%.7 Fifty-eight patients of the 413 identified in this study were treated with gemcitabine, 6.9% showed partial response, 50% remained stable, and 39.7% progressed despite therapy. Median survival was 8.05 months with a hazard ratio (HR) of 0.50 (95% confidence interval 0.35-0.72). Sixteen out of the 58 patients treated with gemcitabine had extrahepatic cholangiocarcinoma. In numerous phase II trials of gemcitabine as a single agent, response rates have ranged from 6-30%, with greater than 50% of treated patients having either a partial response or stable disease. 7-12 Median survival (MS) has ranged from 6.5-14 months in these trials. In 2008, guidelines for CT in biliary tract cancers were published in the Journal of Hepatobiliary and Pancreatic Surgery.13 Seven trials using gemcitabine as a single agent were identified, with response rates ranging from 0-36% and MS ranging from 4.6-14 months. In this article the use of gemcitabine in unresectable cancers of the biliary tract was given a recommendation level C1, meaning that its use may be considered, although there is a lack of high-level evidence.13

The combination of 5-FU or it's oral analog capecitabine and gemcitabine chemotherapy alone (without radiation) in the advanced metastatic setting has improved response rates and median overall survivals from around 10% or 6.1 months to 10-36% and 9.7 to 14 months respectively.13a Based on this data it likely should have synergy if both agents are given concurrently with external beam RT. The combination of continuous 5-FU and gemcitabine with external beam radiation in locally advanced pancreatic cancer has been shown to be safe and resulted in a complete response in 2 patients (6.3%), a partial response in 18 patients (56.3%), with an overall all response rate of 62.5% 13b. Based on this data and the similar dose of external RT therapy it seems reasonable and safe to combine the two agents 5-FU and gemcitabine with RT in advanced cholangiocarcinoma. We chose to use 5-FU rather than oral capecitabine due to occasional problems obtaining prescription coverage for this more expensive alternative and the prior available safety data and our own institutional experience using 5-FU and gemcitabine combination with RT for pancreatic cancer.

Radiation Therapy Data for the use of radiation therapy (RT) alone in the setting of unresectable disease is sparse. In a report from Johns Hopkins, a total of 23 patients were treated with a surgical procedure followed by RT.14 Complete resection was accomplished in 14 of these patients and palliative stenting for 9. Postoperative RT doses ranging from 45-63 Gy delivered by external beam radiation therapy (EBRT) followed by brachytherapy boost or EBRT with cone down boost. RT had no effect on overall survival of patients who had undergone complete resection or on patients who were being treated with palliative intent. Of note, none of the patients in this study were treated with concurrent chemotherapy. The subgroup of patients who were stented and then treated with palliative RT applies to our current investigational study group, and in this subset of patients there was no survival benefit for RT alone.

Chemotherapy and Radiation Therapy Because of the success of combined CT and RT in other gastrointestinal cancers, and the unsuccessful attempts at CT and RT alone, multimodality treatment has been applied to cholangiocarcinoma. There is limited data on the use of EBRT in combination with 5-FU specifically for extrahepatic cholangiocarcinoma. In a retrospective review, Kim et al looked at ≥40 Gy EBRT with concomitant bolus 5-FU (500mg/m2) for the first 3-days of each of two weeks of radiation, followed by monthly maintenance chemo with 5-FU for one year.15 Eighty four patients were included, of which 72 had a gross total resection (47 negative margins, 25 microscopically positive margins) and the remaining 12 had palliative procedures prior to the chemoradiation. The 5-year survival was 31%. Although this trial was specifically looking at postoperative chemoradiotherapy, the subset of patients that did not undergo gross total resection would apply to our study population. The 5-year actuarial survival was 14% overall for this subgroup.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over age 18
2. Intra or extrahepatic cholangiocarcinoma confirmed by biopsy/brushings, biliary aneuploidy demonstrated by FISH, or elevated CA 19-9 greater than 100 ng/mL in the presence of a radiographic malignant stricture
3. Deemed surgically unresectable by a surgical oncologist
4. Malignant disease encompassable within a single radiation field
5. ECOG 0-2
6. Laboratory values: Hemoglobin ≥ 8.0 (can be transfused to attain this value), Granulocytes > 1,500, platelets > 100,000/ul

Exclusion Criteria:

1. Chemotherapy within one month of starting radiation therapy
2. Previous abdominal radiotherapy
3. Uncontrolled infection or severe active comorbid disease
4. Previous malignancy in the past five years, excluding nonmelanoma skin cancers and in situ cervical, bladder or uterine cancer
5. Distant metastatic disease (outside regional lymph nodes)
6. Pregnancy or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Anker, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All participants enrolled.
  Brachytherapy or SBRT (Stereotactic body radiation therapy) : Patients receive 45 Gy (gray) external beam radiation therapy including the primary tumor and regular lymph nodes (25 fractions over 5 weeks). Within 1 month of external beam radiation therapy, patients will have boost treatment of 20 Gy in 4 fractions, via Ir-192 brachytherapy or SBRT (Stereotactic Body Radiation Therapy).
  Fluorouracil (5-FU) : 5-FU Injection,USP. This study uses 350 mg/m2/day days 1-5 each week of radiation therapy
  Gemcitabine
Period: Overall Study
Arm/Group | All Patients
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Toxicity Treated With Gemcitabine Every Two Weeks & 5-FU Given Concurrently With External Beam Radiation Therapy , Followed by Brachytherapy or SBRT Boost.
Time Frame: Toxicity was assessed for each patient over the course of the study treatment and follow-up stage which together lasted 9 months. Only one patient was enrolled.
Measure: Number; unit: participants
Groups:
- All Patients: All participants enrolled.
  Brachytherapy or SBRT (Stereotactic body radiation therapy) :
  Fluorouracil (5-FU) :
  Gemcitabine
Arm/Group | All Patients
Number analyzed (Participants) | 1
participants | 1

2. Secondary Outcome: Evaluate Overall Survival Ratefollowing Gemcitabine and 5-FU With Radiation Therapy in Patients With HCC
Time Frame: 9 months
Population: Trial did not meet accrual goals so analysis was not performed
Arm/Group | All Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Evaluate the Rate at Which Patients With Unresectable Extrahepatic Cholangiocarcinoma Become Resectable Following Gemcitabine and Radiation Therapy.
Time Frame: 9 months
Population: Trial did not meet accrual goals so analysis was not performed
Arm/Group | All Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Evaluate Progression Free Survival Rate Following Gemcitabine and 5-FU With Radiation Therapy in Patients With HCC
Time Frame: 9 months
Population: Trial did not meet accrual goals so analysis was not performed
Arm/Group | All Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Evaluate Tumor Response Rate Following Gemcitabine and 5-FU With Radiation Therapy in Patients With HCC
Time Frame: 9 months.
Population: Trial did not meet accrual goals so analysis was not performed
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Evaluate Local Control Rate Following Gemcitabine and 5-FU With Radiation Therapy in Patients With HCC
Time Frame: 9 months
Population: Trial did not meet accrual goals so analysis was not performed
Arm/Group | All Patients
Number analyzed (Participants) | 0

7. Secondary Outcome: Evaluate Rate of Distant Mets Following Gemcitabine and 5-FU With Radiation Therapy in Patients With HCC
Time Frame: 9 months
Population: Trial did not meet accrual goals so analysis was not performed
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
mucositis (Gastrointestinal disorders) | 1 (1)
Intermittent Nausea (Gastrointestinal disorders) | 1 (1)
Intermittent vomiting (Gastrointestinal disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Intermittent constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes